CLINICAL TRIAL: NCT00313989
Title: Evaluation of Osseo-integration After Placement of Dental Implants With Patients Receiving Radiotherapy for Buccopharyngeal Oncology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/125
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2014-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of implants of patients receiving radiotherapy. (Experimental)
  Interventions: Procedure: Evaluation of the success rate of implants

INTERVENTIONS:
Procedure: Evaluation of the success rate of implants — Evaluation of the success rate of implants

SUMMARY:
Follow up of implants with patients receiving radiotherapy for buccopharyngeal oncology. Implants will be placed 6 weeks before start of the radiotherapy or at least 3 months after the end of the radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving radiotherapy (6 weeks later or at least 3 months before) for buccopharyngeal oncology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Recovering and ingrowing of dental implants | 4 to 6 months
Success rate of dental implants | 4 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be